CLINICAL TRIAL: NCT04176328
Title: An Open-label, Dose-escalation Study to Evaluate the Pharmacokinetics of Inhaled Teicoplanin in Cystic Fibrosis Patients
Brief Title: Open-label, Dose-escalation Study to Evaluate the Pharmacokinetics of Inhaled Teicoplanin in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neupharma Srl (Industry)
Collaborators: Sintesi Research Srl (Industry); Aptuit (Industry); Pari Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-PR-01.2019
Record Dates: First submitted 2019-11-08; First posted 2019-11-25 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Methicillin-resistant Staphylococcus aureus; Teicoplanin
MeSH Terms: conditions — Cystic Fibrosis | interventions — Powders; Solvents; Solutions; Injections; Teicoplanin

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, exploratory, open-label, dose-escalation study evaluating the pharmacokinetics of inhaled Teicoplanin in Cystic Fibrosis patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cystic Fibrosis patients treated with Teicoplanin (Experimental): Hospitalized male and female patients aged ≥ 18 years, suffering of Cystic Fibrosis.
  Interventions: Drug: Teicoplanin Sandoz 200 mg powder and solvent for solution for injection or infusion or oral solution.

INTERVENTIONS:
Drug: Teicoplanin Sandoz 200 mg powder and solvent for solution for injection or infusion or oral solution. — Teicoplanin Sandoz administered by inhalation (aerosol).
  Other Names: Teicoplanin

SUMMARY:
Cystic Fibrosis (CF) is the most common autosomal recessive lethal disorders affecting 1:2.500 newborns among Caucasians. CF patients are peculiarly susceptible to infection and colonization of the respiratory tract with pathogens. In particular, Methicillin-resistant Staphylococcus aureus (MRSA) has become the third most prevalent bacterium in CF in the U.S. and has been increasing in other countries. Apart from the difficulty of treating the infection because of its antimicrobial resistances, MRSA is transmissible between individuals with and without CF. Chronic MRSA infection is associated with worse outcomes, and treatment/eradication is challenging. Antibiotic dosing and choices should be optimized to minimize further resistance and to maximize chances of successful therapy. Yet, MRSA has several mechanisms to escape clearance by the immune system and antibiotic killing. For these reasons, a better understanding of preventive measures and early therapy is of key importance. In consideration of all these assessments there is an emerging consensus that MRSA is an important pathogen in CF rather than simply a marker of severe disease. However, to date there are no guidelines or recommendations on the choice of antibiotics for MRSA in CF. Glycopeptides are an important class of antibiotics active against Gram-positive pathogens. These include teicoplanin and vancomycin, which are currently in widespread use and are active against MRSA. Teicoplanin is often preferred to vancomycin for intravenous treatment because of its better safety profile but its use in MRSA lung infection is limited by its limited lung penetration. Teicoplanin is mainly used for injection/infusion. Inhalation of anti-microbial drugs is a cornerstone in the treatment of patients with CF, since inhaled antibiotics decrease the rate of decline of lung function, improve the quality of life, and reduce the frequency of exacerbations and hospital admissions. It is expected that, using inhalation route, efficacy would be improved and risk of resistance reduced. At present, no antibiotic active against MRSA is available as an inhaled formulation. The objective of this phase I, first-in-man clinical study is to identify the dose providing, after single inhalation administration, a sputum Teicoplanin concentrations exceeding the drug concentration required to inhibit bacterial growth for at least 8 hours, while minimizing the development of resistance.

DETAILED DESCRIPTION:
INTRODUCTION & STATE-OF-ART Cystic Fibrosis (CF) is the most common autosomal recessive lethal disorders affecting 1 in 2.500 newborns among Caucasians. CF lung disease reflects a failure in the capacity of airway epithelia to normally hydrate their surface. Poor hydration of airways surfaces leads to reduced mucociliary clearance, adhesion of mucus to airway surfaces and, ultimately, chronic bacterial infection.

On regard the therapeutic strategy, lung infection in CF was mainly treated with antibiotics, anti-inflammatory medicines, bronchodilators and mucolytics. In addition, patients with cystic fibrosis were often given other types of medicines such as pancreatic enzymes and food supplements. They were also advised to exercise and to have physiotherapy.

Patients with CF are peculiarly susceptible to infection and colonization of the respiratory tract with patho-gens. In particular, methicillin-resistant Staphylococcus aureus (MRSA) has become the third most prevalent bacterium in cystic fibrosis (CF) in the United States and has been increasing in other countries. Apart from the difficulty of treating the infection because of its antimicrobial resistances, MRSA is transmissible between individuals with and without CF.

With increasing survival due to improvements of care, an increased frequency of pulmonary infections with new and resistant pathogens has been identified. In particular, the prevalence of Methicillin-resistant Staphylococcus aureus (MRSA) in respiratory cultures of CF patients has increased over the past decade. MRSA pneumonia is likely to be severe and life threatening, with high mortality, compared with non-MRSA pneumonia.

The impact of MRSA on outcomes in CF is not fully understood. In a large epidemiologic study was shown that lung function decline is more rapid in CF children and adolescents with persistent MRSA compared with those without MRSA. Epidemiologic evidence suggests that persistent infection with MRSA is associated with increased use of intra-venous antibiotics, increased hospitalizations, a faster decline of lung function, as well as shortened life expectancy.

During chronic infection, MRSA shows the adaptive mode of growth, which enhances the bacterias' ability to withstand the immune system and antibiotic therapy. In the setting of chronic infection, however, reduction in bacterial density in sputum and increased clinical stability may be appropriate outcomes.

Chronic MRSA infection is associated with worse outcomes, and treatment/eradication is challenging. Antibiotic dosing and choices should be optimized to minimize further resistance and to maximize chances of successful therapy. Yet, MRSA has several mechanisms to escape clearance by the immune system and antibiotic killing. For these reasons, a better understanding of preventive measures and early therapy is of key importance.

Different approaches have been considered in the prevention and management of MRSA infections among patients with CF. In consideration of all these assessments there is an emerging consensus that MRSA is an important pathogen in CF rather than simply a marker of severe disease. However, to date there are no guidelines or recommendations on the choice of antibiotics for MRSA in CF.

Glycopeptides are an important class of antibiotics active against Gram-positive pathogens. Teicoplanin and vancomycin, are two glycopeptide antibiotics currently in widespread use and are active against MRSA. Teicoplanin susceptibility is considered when minimal inhibition concentration (MIC) is < 2 ug/mL. Teicoplanin is produced by Actynoplanes teichomycietus and acts by inhibition of cell wall synthesis. Teicoplanin is often preferred to vancomycin for intravenous treatment because of its better safety profile but its use in MRSA lung infection is limited by its limited lung penetration. Teicoplanin has been marketed for >20 years in most EU countries. Teicoplanin is mainly used for injection/infusion; the oral route of administration is used only for the treatment of pseudomembranous colitis by Clostridium difficilis.

Inhalation of anti-microbial drugs is a cornerstone in the treatment of patients with CF, by providing high drug concentrations locally in the lung while minimizing systemic exposure and thus the potential for side effects. Nebulized antibiotic therapy directly targets airways and lung parenchyma, thereby resulting in increased local concentrations and hence potentially improving efficacy. In CF, inhaled antibiotics decrease the rate of decline of lung function, improve the quality of life, and reduce the frequency of exacerbations and hospital admissions.

Delivery of nebulized Teicoplanin directly to the bronchial tree may offer improved efficacy. It is expected that, using the inhalation route, lung concentrations will be higher than MICs for most bacteria, improving efficacy and reducing the risk of resistance. At present, no antibiotic active against MRSA is available as an inhaled formulation; vancomycin dry powder for inhalation is currently under clinical investigation in the U.S.A. for the treatment of MRSA lung infection.

SUMMARY OF NON-CLINICAL PHARMACOLOGY Teicoplanin inhibits the growth of susceptible organisms by interfering with cell wall biosynthesis at a site different from that affected by beta-lactams. Specific binding to D-alanyl-D-alanine residues blocks peptidoglycan synthesis. The spectrum of activity of Teicoplanin, like that of vancomycin, is restricted to Gram-positive aerobic and anaerobic bacteria. Teicoplanin is generally more active than vancomycin against streptococci and Gram-positive anaerobes; the two agents exhibit similar activity against S. aureus (including MRSA).

Resistance to Teicoplanin is rare but not unknown. SUMMARY OF CLINICAL DATA In clinical trials, Teicoplanin is associated with fewer side effects than vancomycin, while caution is recommended in the elderly, patients with compromised renal function, pre-existing hearing problems or with a history of allergic reactions to vancomycin. Common adverse reactions (≥1/100 to <1/10) include rash, erythema, pruritis, pain at injections site and pyrexia while less common reactions (≥1/1,000 to <1/100) include leucopenia, thrombocytopenia, eosinophilia, anaphylactic reactions dizziness, headache, phlebitis, bronchospasm, diarrhoea, vomiting, nausea and transient increases in transaminases.

Renal failure has been reported in patients treated with Teicoplanin; patients with renal insufficiency, and/or in those receiving Teicoplanin in conjunction with or sequentially with other medicinal products with known nephrotoxic potential (aminoglycosides, colistin, amphotericin B, cyclosporin, and cisplatin) should be carefully monitored, and should include auditory tests. Since Teicoplanin is mainly excreted by the kidney, the dose of Teicoplanin must be adapted in patients with renal impairment.

As with other glycopeptides, ototoxicity (deafness and tinnitus) has been reported in patients treated with Teicoplanin. Patients who develop signs and symptoms of impaired hearing or disorders of the inner ear during treatment with Teicoplanin should be carefully evaluated and monitored, especially in case of prolonged treatment and in patients with renal insufficiency. Patients receiving Teicoplanin in conjunction with or sequentially with other medicinal products with known neurotoxic/ototoxic potential (amino-glycol¬sides, cyclosporin, cisplatin, furosemide and ethacrynic acid) should be carefully monitored and the benefit of Teicoplanin evaluated if hearing deteriorates.

The safety of Teicoplanin has been confirmed by pharmacovigilance data based on approximately 30 years of use in Gram-positive severe infections. There are no human data concerning the use of inhaled Teicoplanin.

SUMMARY OF CLINICAL PHARMACOKINETICS Teicoplanin is currently administered primarily by the parenteral route (intravenous, IV or intra¬muscular, IM). Following intravenous administration, the disposition kinetics are tri-exponential, and the majority of drug is excreted unchanged by glomerular filtration. In patients with normal renal function, the terminal half-life is 87 h. The volume of distribution at steady-state is 860 mL/kg, clearance is 11.4 mL/h/kg and renal clearance is 8.3 mL/h/kg. Teicoplanin is highly bound in plasma to albumin (fraction unbound = 0.1). The pharmacokinetics are linear over a wide dose range (2 to 26 mg/kg). As expected, clearance is higher in children than in adults, and lower in the elderly, associated with a decrease in glomerular filtration rate with advancing years.

Teicoplanin is not absorbed from the gastrointestinal tract and shows negligible oral bioavailability. After IM administration, the bioavailability of Teicoplanin is 90%. After six daily IM administrations at 200 mg, the mean ± SD maximum Teicoplanin concentration (Cmax) is 12.1 ± 0.9 mg/L and occurs at 2h after administration.

RATIONALE FOR THE STUDY The objective of this phase I, first-in-man clinical study is to identify the dose providing, after single inhalation administration, a sputum Teicoplanin concentrations exceeding the drug concentration required to inhibit bacterial growth for at least 8 hours, while minimizing the development of resistance. To this end, the study is designed with single daily escalating doses in subjects with CF. Up to now, no Teicoplanin product for nebulization has been approved either in EU or U.S.A.. Nevertheless, Teicoplanin containing solutions are often used off-label to manage MRSA lung infections in patients with Cystic Fibrosis, usually with nebulization of 200 mg in 3 ml.

Inhalation by nebulization is a typical topical therapy and its efficacy depends on the physicochemical characteristics of the drug solution and of the nebuliser used to generate the aerosol.

In this trial the first dose has been selected after aerodynamic assessment of nebulised aerosol in accordance with European Pharmacopoeia 9th and USP 28. A starting dose of 150 mg will be most likely well tolerated and possibly able to reach the expected concentration in the target tissue.

On the basis of PK features of Teicoplanin (elimination half-life of the product varies from 100 to 170 hours in blood), of time-dependent killing characteristic, of the mechanism of action and of the expected MIC, an AUC0-12 h of more 300 μg/mL*h in the sputum will be effective in controlling MRSA infection. This value is thus an appropriate end point for a preliminary pilot study after single local administration and will likely allow optimal evaluation of the doses to be applied to test clinical efficacy on the basis of the following considerations:

* Repeated administrations, to be applied in later studies, will produce proportionally higher AUC values than single administration;
* Local ratio between AUC and MIC necessary to achieve killing of MRSA are likely lower than systemic ratio;
* Teicoplanin "off-label" experience is usually based on administration of doses unlikely to produce a AUC0-12 h above 300 μg/mL*h in the sputum.

In conclusion, on the basis of literature data an AUC0-12 h above 300 μg/mL*h in the sputum is achievable within the planned protocol, is likely to be clinically relevant in patients with MRSA lung infection and is likely well tolerated even by patients with chronic lung inflammation as those who will be enrolled in the proposed study.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female patients, aged ≥18 years with a confirmed diagnosis of cystic fibrosis.
2. Patients with body weight ≥50 kg and ≤100 kg
3. Patients with body mass index (BMI) between 18.0 and 30 kg/m2.
4. Patients with FEV1 > 50% of predicted.
5. Patients with regular mucus production due to cystic fibrosis.
6. Patients who are able to understand the nature of the study and willing to comply with the protocol requirements.
7. Patients who have signed written informed consent to participate to the study after risks have been fully explained.

EXCLUSION CRITERIA:

1. Patients treated with nebulized antibiotics within 14 days or mucolytic agents, hypertonic saline solution within 48 hours before administration of the Investigational Product or during the study.
2. Patients with medical history of hemoptysis (> 300 cc in 30 days).
3. Patients with decreased liver function (AST or ALT > 3 times higher in comparison to reference values).
4. Patients with eGFR < 60 mL/min/1.73 m2
5. Patients on the waiting list for lung transplantation.
6. Patients with known or suspected allergy or hypersensitivity to glycopeptides.
7. Patients treated with Teicoplanin for inhalation and systemic within 4 weeks before each dosing occasion.
8. Patients with known episodes of bronchoconstriction after drug inhalation.
9. Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment.
10. Female patients who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical study and for one months later.
11. Female patients of childbearing age (less than 24 months after the last menstrual cycle) who do not use adequate contraception. * * Methods at low risk of contraceptive failure (less than 1% per year) when used consistently, including: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), some intra-uterine devices, abstinence or vasectomized partner. Contraception should be maintained until 1 month after the last visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Concentration of Teicoplanin in the sputum of CF patients treated with inhaled Teicoplanin. | Change occurring from pre-inhalation (0 hours) to the following time points: after 0.5 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 30 hours, 48 hours from each inhalation.
  Measurement of the concentration (expressed as mg/L) of Teicoplanin in the sputum of patients suffering of Cystic Fibrosis after a single inhalation of 150 mg at scheduled time points after first inhalation: 0 hours, 0.5 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 30 hours, 48 hours. In case a value of sputum AUC0-12 h above 300 μg/mL*h will not be achieved with the first dosage inhalation of Teicoplanin, up to two additional inhalations with different dosages will be foreseen and the same time points will be measured for subsequent inhalations. In addition, the inhalation of Teicoplanin with the maximum (300 mg) dosage foreseen by study protocol is expected for all patients aiming to confirm the optimal intermediate dosage tested during the dose-escalation process.

SECONDARY OUTCOMES:
Concentration of Teicoplanin in the blood of CF patients treated with inhaled Teicoplanin. | Change occurring from pre-inhalation (0 hours) to the following time points: after 0.5 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours from each inhalation.
  Measurement of the concentration (expressed as mg/L) of Teicoplanin in the blood of patients suffering of Cystic Fibrosis after a single inhalation of 150 mg at scheduled time points after first inhalation: 0 hours, 0.5 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours. In case a value of sputum AUC0-12 h above 300 μg/mL*h will not be achieved with the first dosage inhalation of Teicoplanin, up to two additional inhalations with different dosages will be foreseen and the same time points will be measured for subsequent inhalations. In addition, the inhalation of Teicoplanin with the maximum (300 mg) dosage foreseen by study protocol is expected for all patients aiming to confirm the optimal intermediate dosage tested during the dose-escalation process.
Concentration of Teicoplanin in the urine of CF patients treated with inhaled Teicoplanin. | Change occurring from pre-inhalation (0 hours) to the following time points: during the intervals 0-4 hours, 4-12 hours, 12-24 hours from each inhalation + after 48 hours from inhalation.
  Measurement of the concentration (expressed as mg/L) of Teicoplanin in the urine of patients suffering of Cystic Fibrosis after a single inhalation of 150 mg at scheduled time intervals after first inhalation: 0 h, 0 - 4 h, 4 - 12 h, 12 - 24 h and after 48 hours from inhalation. In case a value of sputum AUC0-12 h above 300 μg/mL*h will not be achieved with the first dosage inhalation of Teicoplanin, up to two additional inhalations with different dosages will be foreseen and the same time intervals will be measured for subsequent inhalations. In addition, the inhalation of Teicoplanin with the maximum (300 mg) dosage foreseen by study protocol is expected for all patients aiming to confirm the optimal intermediate dosage tested during the dose-escalation process.
Comparison between concentrations of Teicoplanin in the sputum, blood and urine of CF patients treated with inhaled Teicoplanin. | During each inhalation visit throughout study period, an average of 3 months per patient.
  Comparison between the concentration (expressed as mg/L) of Teicoplanin measured in the sputum, blood and urine of patients suffering of Cystic Fibrosis after a single inhalation of 150 mg versus additional dosages of Teicoplanin (including the maximum dosage tested).
Percentage of change of FEV1 value (by means of Spirometry test) in comparison to baseline (pre-inhalation) in CF patients treated with inhaled Teicoplanin (as part of Tolerability outcome). | 30 minutes pre-inhalation + after 30 minutes, 60 minutes and 120 minutes (if needed) from each inhalation.
  Measurement of any changes (as percent) in the Forced Expiratory Volume in the 1st second (FEV1) measured 30 minutes before and 30 and 60 minutes after a single inhalation of 150 mg of inhaled Teicoplanin. In case of FEV1 reduction > 5% in comparison to baseline the FEV1 will be measured also after 120 minutes from inhalation.
Percentage of change of blood oxigen saturation value (by means of Pulse Oximetry test) in comparison to baseline (pre-inhalation) in CF patients treated with inhaled Teicoplanin (as part of Tolerability outcome). | 30 minutes pre-inhalation + after 30 minutes and 4 hours from each inhalation.
  Measurement of any changes (as percent) in the blood oxigen saturation measured 30 minutes before and 30 minutes + 4 hours after a single inhalation of 150 mg of inhaled Teicoplanin.
Rate and characterization of adverse events occurring to CF patients treated with inhaled Teicoplanin (as part of Safety outcome). | During the entire study period, an average of 3 months per patient.
  Evaluation of the number, rate and characteristics of the adverse events occurring to CF patients treated with inhaled Teicoplanin, as recorded in the Case Report Form. Any adverse events occurring during the inhalation visits will be also evaluated from a Tolerability point of view.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Paiola, MD, Principal Investigator — U.O.C. Fibrosi Cistica - Azienda Ospedaliera Universitaria Integrata di Verona
Locations (1):
- Centro Ricerche Cliniche di Verona - Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ratjen F, Doring G. Cystic fibrosis. Lancet. 2003 Feb 22;361(9358):681-9. doi: 10.1016/S0140-6736(03)12567-6. PMID 12606185
- [Background] Elborn JS. Cystic fibrosis. Lancet. 2016 Nov 19;388(10059):2519-2531. doi: 10.1016/S0140-6736(16)00576-6. Epub 2016 Apr 29. PMID 27140670
- [Background] Ratjen F. Diagnosing and managing infection in CF. Paediatr Respir Rev. 2006;7 Suppl 1:S151-3. doi: 10.1016/j.prrv.2006.04.217. Epub 2006 Jun 6. PMID 16798546
- [Background] Huang YJ, LiPuma JJ. The Microbiome in Cystic Fibrosis. Clin Chest Med. 2016 Mar;37(1):59-67. doi: 10.1016/j.ccm.2015.10.003. Epub 2015 Dec 23. PMID 26857768
- [Background] Burns JL, Gibson RL, McNamara S, Yim D, Emerson J, Rosenfeld M, Hiatt P, McCoy K, Castile R, Smith AL, Ramsey BW. Longitudinal assessment of Pseudomonas aeruginosa in young children with cystic fibrosis. J Infect Dis. 2001 Feb 1;183(3):444-52. doi: 10.1086/318075. Epub 2000 Dec 27. PMID 11133376
- [Background] Frederiksen B, Koch C, Hoiby N. Changing epidemiology of Pseudomonas aeruginosa infection in Danish cystic fibrosis patients (1974-1995). Pediatr Pulmonol. 1999 Sep;28(3):159-66. doi: 10.1002/(sici)1099-0496(199909)28:33.0.co;2-1. PMID 10495331
- [Background] Emerson J, Rosenfeld M, McNamara S, Ramsey B, Gibson RL. Pseudomonas aeruginosa and other predictors of mortality and morbidity in young children with cystic fibrosis. Pediatr Pulmonol. 2002 Aug;34(2):91-100. doi: 10.1002/ppul.10127. PMID 12112774
- [Background] Henry RL, Mellis CM, Petrovic L. Mucoid Pseudomonas aeruginosa is a marker of poor survival in cystic fibrosis. Pediatr Pulmonol. 1992 Mar;12(3):158-61. doi: 10.1002/ppul.1950120306. PMID 1641272
- [Background] Ballmann M, Rabsch P, von der Hardt H. Long-term follow up of changes in FEV1 and treatment intensity during Pseudomonas aeruginosa colonisation in patients with cystic fibrosis. Thorax. 1998 Sep;53(9):732-7. doi: 10.1136/thx.53.9.732. PMID 10319054
- [Background] Waters V. New treatments for emerging cystic fibrosis pathogens other than Pseudomonas. Curr Pharm Des. 2012;18(5):696-725. doi: 10.2174/138161212799315939. PMID 22229574
- [Background] Parkins MD, Floto RA. Emerging bacterial pathogens and changing concepts of bacterial pathogenesis in cystic fibrosis. J Cyst Fibros. 2015 May;14(3):293-304. doi: 10.1016/j.jcf.2015.03.012. Epub 2015 Apr 14. PMID 25881770
- [Background] Vanderhelst E, De Meirleir L, Verbanck S, Pierard D, Vincken W, Malfroot A. Prevalence and impact on FEV(1) decline of chronic methicillin-resistant Staphylococcus aureus (MRSA) colonization in patients with cystic fibrosis. A single-center, case control study of 165 patients. J Cyst Fibros. 2012 Jan;11(1):2-7. doi: 10.1016/j.jcf.2011.08.006. Epub 2011 Sep 9. PMID 21907637
- [Background] Dasenbrook EC, Merlo CA, Diener-West M, Lechtzin N, Boyle MP. Persistent methicillin-resistant Staphylococcus aureus and rate of FEV1 decline in cystic fibrosis. Am J Respir Crit Care Med. 2008 Oct 15;178(8):814-21. doi: 10.1164/rccm.200802-327OC. Epub 2008 Jul 31. PMID 18669817
- [Background] Boxerbaum B, Jacobs MR, Cechner RL. Prevalence and significance of methicillin-resistant Staphylococcus aureus in patients with cystic fibrosis. Pediatr Pulmonol. 1988;4(3):159-63. doi: 10.1002/ppul.1950040307. PMID 3259692
- [Background] Miall LS, McGinley NT, Brownlee KG, Conway SP. Methicillin resistant Staphylococcus aureus (MRSA) infection in cystic fibrosis. Arch Dis Child. 2001 Feb;84(2):160-2. doi: 10.1136/adc.84.2.160. PMID 11159295
- [Background] Goodrich JS, Sutton-Shields TN, Kerr A, Wedd JP, Miller MB, Gilligan PH. Prevalence of community-associated methicillin-resistant Staphylococcus aureus in patients with cystic fibrosis. J Clin Microbiol. 2009 Apr;47(4):1231-3. doi: 10.1128/JCM.00255-09. Epub 2009 Feb 18. PMID 19225098
- [Background] Harik NS, Com G, Tang X, Melguizo Castro M, Stemper ME, Carroll JL. Clinical characteristics and epidemiology of methicillin-resistant Staphylococcus aureus (MRSA) in children with cystic fibrosis from a center with a high MRSA prevalence. Am J Infect Control. 2016 Apr 1;44(4):409-15. doi: 10.1016/j.ajic.2015.10.015. Epub 2015 Dec 9. PMID 26684366
- [Background] Goss CH, Muhlebach MS. Review: Staphylococcus aureus and MRSA in cystic fibrosis. J Cyst Fibros. 2011 Sep;10(5):298-306. doi: 10.1016/j.jcf.2011.06.002. Epub 2011 Jun 29. PMID 21719362
- [Background] Lo DK, Hurley MN, Muhlebach MS, Smyth AR. Interventions for the eradication of meticillin-resistant Staphylococcus aureus (MRSA) in people with cystic fibrosis. Cochrane Database Syst Rev. 2015 Feb 24;(2):CD009650. doi: 10.1002/14651858.CD009650.pub3. PMID 25927091
- [Background] Schreiber MP, Chan CM, Shorr AF. Resistant pathogens in nonnosocomial pneumonia and respiratory failure: is it time to refine the definition of health-care-associated pneumonia? Chest. 2010 Jun;137(6):1283-8. doi: 10.1378/chest.09-2434. Epub 2010 Feb 12. PMID 20154075
- [Background] Hidron AI, Low CE, Honig EG, Blumberg HM. Emergence of community-acquired meticillin-resistant Staphylococcus aureus strain USA300 as a cause of necrotising community-onset pneumonia. Lancet Infect Dis. 2009 Jun;9(6):384-92. doi: 10.1016/S1473-3099(09)70133-1. PMID 19467478
- [Background] Dasenbrook EC, Checkley W, Merlo CA, Konstan MW, Lechtzin N, Boyle MP. Association between respiratory tract methicillin-resistant Staphylococcus aureus and survival in cystic fibrosis. JAMA. 2010 Jun 16;303(23):2386-92. doi: 10.1001/jama.2010.791. PMID 20551409
- [Background] Gur M, Spinelli E, Tridello G, Baltieri S, Pinali L, Montemezzi S, Bentur L, Assael BM. Chest computed tomography scores in patients with cystic fibrosis colonized with methicillin-resistant Staphylococcus aureus. Clin Respir J. 2018 Feb;12(2):779-785. doi: 10.1111/crj.12594. Epub 2017 May 4. PMID 27925453
- [Background] Solis A, Brown D, Hughes J, Van Saene HK, Heaf DP. Methicillin-resistant Staphylococcus aureus in children with cystic fibrosis: An eradication protocol. Pediatr Pulmonol. 2003 Sep;36(3):189-95. doi: 10.1002/ppul.10231. PMID 12910579
- [Background] Muhlebach MS. Methicillin-resistant Staphylococcus aureus in cystic fibrosis: how should it be managed? Curr Opin Pulm Med. 2017 Nov;23(6):544-550. doi: 10.1097/MCP.0000000000000422. PMID 28796008
- [Background] Dolce D, Neri S, Grisotto L, Campana S, Ravenni N, Miselli F, Camera E, Zavataro L, Braggion C, Fiscarelli EV, Lucidi V, Cariani L, Girelli D, Faelli N, Colombo C, Lucanto C, Lombardo M, Magazzu G, Tosco A, Raia V, Manara S, Pasolli E, Armanini F, Segata N, Biggeri A, Taccetti G. Methicillin-resistant Staphylococcus aureus eradication in cystic fibrosis patients: A randomized multicenter study. PLoS One. 2019 Mar 22;14(3):e0213497. doi: 10.1371/journal.pone.0213497. eCollection 2019. PMID 30901344
- [Background] Reynolds PE. Structure, biochemistry and mechanism of action of glycopeptide antibiotics. Eur J Clin Microbiol Infect Dis. 1989 Nov;8(11):943-50. doi: 10.1007/BF01967563. PMID 2532132
- [Background] Ramos-Martin V, Johnson A, McEntee L, Farrington N, Padmore K, Cojutti P, Pea F, Neely MN, Hope WW. Pharmacodynamics of teicoplanin against MRSA. J Antimicrob Chemother. 2017 Dec 1;72(12):3382-3389. doi: 10.1093/jac/dkx289. PMID 28962026
- [Background] Cavalcanti AB, Goncalves AR, Almeida CS, Bugano DD, Silva E. Teicoplanin versus vancomycin for proven or suspected infection. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD007022. doi: 10.1002/14651858.CD007022.pub2. PMID 20556772
- [Background] Wilson AP. Clinical pharmacokinetics of teicoplanin. Clin Pharmacokinet. 2000 Sep;39(3):167-83. doi: 10.2165/00003088-200039030-00001. PMID 11020133
- [Background] Quon BS, Goss CH, Ramsey BW. Inhaled antibiotics for lower airway infections. Ann Am Thorac Soc. 2014 Mar;11(3):425-34. doi: 10.1513/AnnalsATS.201311-395FR. PMID 24673698
- [Background] Greenwood D. Microbiological properties of teicoplanin. J Antimicrob Chemother. 1988 Jan;21 Suppl A:1-13. doi: 10.1093/jac/21.suppl_a.1. PMID 2965119
- [Background] Sipahi OR, Arda B, Yurtseven T, Sipahi H, Ozgiray E, Suntur BM, Ulusoy S. Vancomycin versus teicoplanin in the therapy of experimental methicillin-resistant Staphylococcus aureus (MRSA) meningitis. Int J Antimicrob Agents. 2005 Nov;26(5):412-5. doi: 10.1016/j.ijantimicag.2005.08.011. Epub 2005 Oct 10. PMID 16221540
- [Background] Parenti F. Structure and mechanism of action of teicoplanin. J Hosp Infect. 1986 Mar;7 Suppl A:79-83. doi: 10.1016/0195-6701(86)90011-3. PMID 2871101
- [Background] Svetitsky S, Leibovici L, Paul M. Comparative efficacy and safety of vancomycin versus teicoplanin: systematic review and meta-analysis. Antimicrob Agents Chemother. 2009 Oct;53(10):4069-79. doi: 10.1128/AAC.00341-09. Epub 2009 Jul 13. PMID 19596875
- [Background] Beltrametti F, Consolandi A, Carrano L, Bagatin F, Rossi R, Leoni L, Zennaro E, Selva E, Marinelli F. Resistance to glycopeptide antibiotics in the teicoplanin producer is mediated by van gene homologue expression directing the synthesis of a modified cell wall peptidoglycan. Antimicrob Agents Chemother. 2007 Apr;51(4):1135-41. doi: 10.1128/AAC.01071-06. Epub 2007 Jan 12. PMID 17220405
- [Background] Mercier E, Darrouzain F, Montharu J, Guillon A, Diot P, Paintaud G, Vecellio L. Lung and serum teicoplanin concentration after aerosol and intravenous administration in a rat model. J Aerosol Med Pulm Drug Deliv. 2014 Aug;27(4):306-12. doi: 10.1089/jamp.2013.1060. Epub 2013 Dec 9. PMID 24320618
- [Background] Guillon A, Mercier E, Lanotte P, Haguenoer E, Darrouzain F, Barc C, Sarradin P, Si-Tahar M, Heuze-Vourc'h N, Diot P, Vecellio L. Aerosol Route to Administer Teicoplanin in Mechanical Ventilation: In Vitro Study, Lung Deposition and Pharmacokinetic Analyses in Pigs. J Aerosol Med Pulm Drug Deliv. 2015 Aug;28(4):290-8. doi: 10.1089/jamp.2014.1164. Epub 2015 Jan 23. PMID 25616054
- [Background] Matsumoto K, Watanabe E, Kanazawa N, Fukamizu T, Shigemi A, Yokoyama Y, Ikawa K, Morikawa N, Takeda Y. Pharmacokinetic/pharmacodynamic analysis of teicoplanin in patients with MRSA infections. Clin Pharmacol. 2016 Mar 30;8:15-8. doi: 10.2147/CPAA.S96143. eCollection 2016. PMID 27099534
- [Background] Cystic Fibrosis foundation Patient Registry: Annual Data Report 2015
- [Background] Teicoplanin Sandoz powder and solvent for solution 200 mg in 3 mL - Summary of the product characteristics
- [Background] Denton M. Re: "Methicillin-resistant Staphylococcus aureus in children with cystic fibrosis: an eradication protocol" Solis et al. (Pediatr Pulmonol 2003;36: 189-195). Pediatr Pulmonol. 2004 Sep;38(3):272-3. doi: 10.1002/ppul.20070. No abstract available. PMID 15274111